CLINICAL TRIAL: NCT00860418
Title: Pediatric Asthma Alert Intervention for Minority Children
Brief Title: Pediatric Asthma Alert Intervention for Minority Children With Asthma
Acronym: PAAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Arlene M. Butz, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NR010546
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: asthma; feedback; anti-inflammatory; ED visits
MeSH Terms: conditions — Asthma | interventions — Nurses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard asthma education delivered during 2 home visits by a nurse.
  Interventions: Behavioral: Standard asthma education
- 2 PAAL (Experimental): PAAL
  Interventions: Behavioral: Pediatric Asthma Alert (PAAL)

INTERVENTIONS:
Behavioral: Pediatric Asthma Alert (PAAL) — Asthma nurse conducts 2 home visits and accompanies the child to primary care provider visit after ED visits
  Other Names: Pediatric Asthma Alert Leader (Nurse)
  Arms: 2 PAAL
Behavioral: Standard asthma education — Standard asthma education during 2 home visits.
  Other Names: Asthma Education
  Arms: 1

SUMMARY:
Young inner-city children with asthma have the highest emergency department (ED) visit rates. Relying on the emergency department for asthma care can be a dangerous sign of poorly controlled asthma. This research will focus on whether having a specialized asthma nurse join the family at a child's doctor visit after an ED visit for asthma to make sure the child and parent keep the follow-up appointment and have the nurse remind the child's doctor to prescribe preventive asthma medicines and an asthma action plan for home (PAAL intervention) will result in young children with asthma having fewer days with wheezing and cough.

The investigators hypothesize that:

1. Significantly more children receiving the PAAL intervention will attend greater than 2 non-urgent visits and greater than 6 refills for the child's anti-inflammatory medications over 12 months when compared to children in the control or standard asthma education group.
2. Children in the PAAL intervention group will experience less morbidity and caregivers will experience increased quality of life compared to children in the control of standard asthma education group.

DETAILED DESCRIPTION:
Asthma is the number one cause of pediatric emergency department (ED) visits in young children and results in a significant economic impact on society and use of health resources. Reliance on the ED for asthma care is not only costly but it is also a dangerous index of poorly controlled asthma. Recent updated national asthma guidelines recommend daily inhaled corticosteroids (ICS) as the cornerstone of treatment for patients with persistent asthma. When properly used ICS prevent exacerbations, ED visits and hospitalizations and maintain asthma control. However, > 50% of inner city minority children with asthma do not receive or use recommended anti-inflammatory preventive medications. In fact, many children encounter repeated ED visits with no provision of appropriate preventive medications or other components of guideline-based preventive care because of inconsistent follow-up with their primary care provider (PCP). The overall goal of this study is to evaluate whether a standardized caregiver and physician prompting intervention, Pediatric Asthma Alert Leader (PAAL), can improve guideline-based preventive asthma care including increased anti-inflammatory use and preventive PCP visits in children with frequent ED visits. This study builds on the experience with our parent-child-PCP communication intervention ("Improving Asthma Communication in Minority Families", ACE) in which we found that teaching parent and child asthma communication skills resulted in increased anti-inflammatory medication use at 6 months for children with persistent asthma. However, the beneficial effects of this intervention were seen primarily when caregivers and children were reminded by the nurse interventionist to relay specific health information to the PCP. Furthermore, the intervention was not associated with decreased ED visits or appropriate PCP follow-up to sustain preventive care. The proposed PAAL intervention has the potential to substantially improve care for children at highest risk for asthma morbidity and we propose to establish (1) whether the positive effects of the ACE study can be replicated in a specific group of high-risk children with repeat ED visits; 2) whether the effects of the intervention can be enhanced by incorporating consistent clinician prompting to assure the provision of each component of guideline-based asthma care (ICS use, asthma action plan, and sustaining regular follow-up care to monitor asthma control); and 3)whether families not achieving optimal care will respond to a more intensive tiered intervention. We propose a caregiver and clinician prompting/feedback intervention using a pediatric asthma alert leader (PAAL) nurse to 1) organize and relay critical, individualized child health information from the ED and home setting to the PCP in a feedback letter, 2) ensure child and caregiver attendance at the follow-up visit with the PCP and 3) empower the family and prompt the PCP for guideline-based treatment decisions at the PCP visit. We hypothesize that the PAAL intervention will improve preventive care and reduce morbidity and health care costs for high-risk children with asthma compared to a Standard Asthma Education (SAE) control group.

ELIGIBILITY:
Inclusion Criteria:

All 6 criteria must be met:

1. Physician-diagnosed asthma (based on caregiver report with validation from the child's physician)
2. > 2 ED visits or > 1 hospitalization for asthma within past 12 months
3. Mild persistent to severe persistent asthma based on NHLBI guidelines criteria (7-9) having any 1 of the following:

   * An average of > 2 days per week of asthma symptoms
   * > 2 days per week with rescue medication use (albuterol, xopenex) OR
   * > 2 days per month of nighttime symptoms
4. Age > 3 and < 10 years
5. Reside in Baltimore Metropolitan area
6. Not currently participating in another asthma study or sibling enrolled in PAAL study

Exclusion Criteria:

1. Inability to speak and understand English
2. No access to a working phone or alternate phone for follow-up surveys
3. Co-morbid respiratory condition including cystic fibrosis, chronic lung disease (BPD), lung cancer, tracheostomy that could interfere with the assessment of asthma-related outcome measures.
4. Children residing in foster care or where consent cannot be obtained from a legal guardian.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of primary care appointments kept over 12 months | 12 months

SECONDARY OUTCOMES:
Number of refills for anti-inflammatory medications prescribed over 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arlene M Butz, ScD, RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Bellin MH, Margolis RH, Whitney L, Osteen P, Thompson A, Butz AM. Violence Exposure, Child Asthma Morbidity, and Maternal Depressive Symptoms: A Longitudinal Analysis of Cumulative Risk. J Health Care Poor Underserved. 2022;33(1):47-66. doi: 10.1353/hpu.2022.0006. PMID 35153205
- [Derived] Bellin MH, Osteen P, Kub J, Bollinger ME, Tsoukleris M, Chaikind L, Butz AM. Stress and Quality of Life in Urban Caregivers of Children With Poorly Controlled Asthma: A Longitudinal Analysis. J Pediatr Health Care. 2015 Nov-Dec;29(6):536-46. doi: 10.1016/j.pedhc.2015.04.018. Epub 2015 May 30. PMID 26036621
- [Derived] Butz AM, Halterman J, Bellin M, Kub J, Tsoukleris M, Frick KD, Thompson RE, Land C, Bollinger ME. Improving preventive care in high risk children with asthma: lessons learned. J Asthma. 2014 Jun;51(5):498-507. doi: 10.3109/02770903.2014.892608. Epub 2014 Feb 27. PMID 24517110
- [Derived] Butz AM, Halterman JS, Bellin M, Kub J, Frick KD, Lewis-Land C, Walker J, Donithan M, Tsoukleris M, Bollinger ME. Factors associated with completion of a behavioral intervention for caregivers of urban children with asthma. J Asthma. 2012 Nov;49(9):977-88. doi: 10.3109/02770903.2012.721435. Epub 2012 Sep 19. PMID 22991952